CLINICAL TRIAL: NCT00471822
Title: An Evaluation of Streptococcus Pneumoniae Serotype Carriage Rate for Nasopharyngeal Carriage in Taiwanese Children Attending Pediatric Clinics in Hospitals, Day Care Centers, or Kindergartens
Brief Title: Nasopharyngeal Streptococcus Pneumoniae Carriage
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0887X-101849; B1841034
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-09

CONDITIONS: Streptococcus Pneumoniae Infections
Keywords: Streptococcus pneumoniae nasopharyngeal carriage
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Primary Objective: Evaluation of the

- Carriage rate of Streptococcus pneumoniae in the nasopharynx of children

Secondary Objective:

* Carriage rate and distribution of Streptococcus pneumoniae serotypes
* Estimation of prevalence rate of antibiotic-resistant Streptococcus pneumoniae strains
* Distribution of Staphylococcus aureus strain
* The influence of risk factors in the Streptococcus pneumoniae carriage rate in children

ELIGIBILITY:
Inclusion Criteria:

1. Children aged between 2 months and 5 years attending pediatric clinics in hospitals, day care centers or kindergartens.
2. Informed consent obtained from parents or legal guardian.

Exclusion Criteria:

1. Children younger than 2 months of age.
2. Children with following serious diseases: immunological disease, neoplastic disease, renal, cardiac or hematological disease, bronchodysplasia, Down's syndrome.

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects aged between 2 months and 5 years attending pediatric clinics in hospitals, daycare centers, and kindergartens
Sampling Method: Non-Probability Sample
Enrollment: 9707 (Actual)
Dates: Start 2005-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Taoyuan District, Taiwan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0887X-101849&StudyName=Nasopharyngeal%20Streptococcus%20Pneumoniae%20Carriage

RESULTS

PARTICIPANT FLOW:
Groups:
- All Potential Carriers: Participants with age range of 2 months to 5 years at pediatric clinics in hospitals, day care centers or kindergartens, with potential carriage of streptococcus pneumoniae strains.
Period: Overall Study
Arm/Group | All Potential Carriers
Started | 9707
Treated | 9705
Completed | 9705
Not Completed | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | All Potential Carriers
Number analyzed (Participants) | 9705
Age Continuous [Mean (Standard Deviation); unit: Years] | 2.05 (1.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4429
  Male | 5276

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Carriage of Streptococcus Pneumoniae in Nasopharynx
Description: Swab cultures obtained from the nasopharynx of participants were tested for the presence of streptococcus pneumoniae strains.
Time Frame: Day 1
Population: Evaluable population included all the participants who met inclusion and exclusion criteria for the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | All Potential Carriers
Number analyzed (Participants) | 9705
Percentage of Participants | 12.6

2. Secondary Outcome: Serotype Distribution of Streptococcus Pneumoniae Isolates
Description: Streptococcus pneumoniae in swab culture of nasopharynx were serotyped. The assessment included 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, 33F, non-vaccine, non-typable and missing serotypes. Percentage of participants under different vaccine serotypes in identified isolates of streptococcus pneumonia are reported.
Time Frame: Day 1
Population: Evaluable population included all the participants who met inclusion and exclusion criteria for the study. Here, 'N' (number of participants analyzed) signifies those participants who were carrier of streptococcus pneumoniae in nasopharynx.
Measure: Number; unit: Percentage of Carrier Participants
Arm/Group | All Potential Carriers
Number analyzed (Participants) | 1225
Percentage of Carrier Participants
  1 | 0.00
  2 | 0.08
  3 | 0.98
  4 | 0.00
  5 | 0.00
  6B | 18.04
  7F | 0.00
  8 | 0.41
  9N | 0.08
  9V | 0.41
  10A | 0.16
  11A | 0.24
  12F | 0.00
  14 | 6.37
  15B | 5.63
  17F | 0.00
  18C | 0.16
  19A | 1.88
  19F | 17.47
  20 | 0.00
  22F | 0.16
  23F | 11.59
  33F | 0.00
  Non-vaccine serotype | 21.80
  Non-typable | 12.33
  Missing | 2.20

3. Secondary Outcome: Antibiotic-Resistant Streptococcus Pneumoniae Strains
Description: Antibiotic resistance is defined as in vitro inhibition of a particular bacterial strain by a concentration of the drug associated with high likelihood of therapeutic failure. Antibiotic resistance for streptococcus pneumoniae was assessed against Penicillin, Cefotaxime, Levofloxacin, Erythromycin and combination of Trimethoprim with sulfamethoxazole. The standard breakpoint value (microbial growth inhibition zone) for Penicillin, Cefotaxime, Levofloxacin, Erythromycin and combination of Trimethoprim with sulfamethoxazole was not more than 8, 4, 13, 15 and 15 millimeter (mm) respectively. Percentage of participants with antibiotic-resistant streptococcus pneumoniae strains are reported. The same participant may have streptococcus pneumoniae strains which is resistance to more than one antibiotic.
Time Frame: Day 1
Population: as for outcome 2
Measure: Number; unit: Percentage of Carrier Participants
Arm/Group | All Potential Carriers
Number analyzed (Participants) | 1225
Percentage of Carrier Participants
  Penicillin | 0.65
  Cefotaxime | 3.51
  Levofloxacin | 1.47
  Erythromycin | 95.43
  Trimethoprim-sulfamethoxazole | 76.00

4. Secondary Outcome: Percentage of Participants With Carriage of Staphylococcus Aureus in Nostril
Description: Swab cultures obtained from the nostril of participants were tested for the presence of Staphylococcus aureus strains.
Time Frame: Day 1
Population: Evaluable population included all participants who met inclusion and exclusion criteria for the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | All Potential Carriers
Number analyzed (Participants) | 9705
Percentage of Participants | 25.9

5. Secondary Outcome: Percentage of Participants With Carriage of Streptococcus Pneumoniae Based on Risk Factors
Description: Participants for carriage of streptococcus pneumoniae were analyzed with respect to various risk factors which included number of bathrooms, number of siblings in the family (multiple siblings), size of the house in meter square (house area), frequency of hand wash in a day, bed sharing, smoking by family member, child breast feeding (breast milk practice), daycare attendance, vaccination for flu and pneumococcus, history of otitis media and upper respiratory infection (URI), antibiotic use and influenza virus infection.
Time Frame: Day 1
Population: Evaluable population included all the participants who met inclusion and exclusion criteria for the study. 'n' signifies those participants who were evaluated for the respective risk factor.
Measure: Number; unit: Percentage of Participants
Arm/Group | All Potential Carriers
Number analyzed (Participants) | 9705
Percentage of Participants
  Bathroom : Less than or equal to (<=) 2 (n=6061) | 12.6
  Bathroom : Greater than (>) 2 (n=3644) | 12.7
  House area : <=50 (n=5698) | 12.5
  House area : >50 (n=4007) | 12.9
  Multiple siblings : >1 (n=6383) | 14.9
  Multiple siblings : Only 1 (n=3320) | 8.3
  Frequency of hand wash : Less than (<) 4 (n=2646) | 9.1
  Frequency of hand wash : 4 to 8 (n=5276) | 14.2
  Frequency of hand wash : >8 (n=1783) | 13.1
  Bed sharing : Yes (n=8689) | 12.9
  Bed sharing : No (n=1016) | 10.1
  Family member smoking : Yes (n=4546) | 13.8
  Family member smoking : No (n=5159) | 11.6
  Breast milk practice : Yes (n=7000) | 12.2
  Breast milk practice : No (n=2705) | 13.6
  Daycare attendance : Yes (n=1783) | 25.4
  Daycare attendance : No (n=7922) | 9.8
  Flu vaccine : Yes (n=3993) | 13.7
  Flu vaccine : No (n=5712) | 11.9
  Pneumoccal vaccine : Yes (n=2225) | 9.8
  Pneumoccal vaccine : No (n=7480) | 13.4
  Otitis media : Yes (n=894) | 21.6
  Otitis media : No (n=8811) | 11.7
  URI in last 2 weeks : Yes (n=2940) | 19.5
  URI in last 2 weeks : No (n=6765) | 9.6
  Antibiotic use : Yes (n=574) | 22.1
  Antibiotic use : No (n=9131) | 12.0
  Influenza virus infection : Yes (n=21) | 28.6
  Influenza virus infection : No (n=9684) | 12.6

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | All Potential Carriers
Serious Adverse Events (participants affected / at risk) | 1/9705
Other Adverse Events (participants affected / at risk) | 359/9705
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Potential Carriers (N=9705)
Bronchiolitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Potential Carriers (N=9705)
Diarrhoea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 2
Pyrexia (General disorders) | 117
Bronchiolitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpangina (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 46
Otitis media acute (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Injury (Injury, poisoning and procedural complications) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 60
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 115
Sneezing (Respiratory, thoracic and mediastinal disorders) | 25
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 7
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.